CLINICAL TRIAL: NCT00992901
Title: Hormonal and Neural Control of Insulin Secretion Following Gastric Bypass Surgery
Brief Title: Role of Neural and Hormonal Regulation Factors on Insulin Secretion After Gastric Bypass Surgery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18-070H; DK083554 (Other Grant/Funding Number: NIDDK)
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Post Bariatricsurgery; Hypoglycemia
Keywords: gastric bypass surgery; glucose tolerance; Insulin response to meal ingestion; Gut hormone and neural response to meal ingestion
MeSH Terms: conditions — Hypoglycemia | interventions — exendin (9-39); Atropine; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exendin-(9-39) (Experimental): To evaluate the role of GLP-1 signaling in glucose tolerance and insulin secretion
  Interventions: Drug: Exendin-(9-39)
- atropine (Experimental): To evaluate the effect of neural activation on insulin secretion and glucose metabolism
  Interventions: Drug: Atropine
- GLP-1 and GIP (Experimental): to evaluate the beta-cell sensitivity to different doses of exogenous gut hormones
  Interventions: Drug: GLP-1 and GIP

INTERVENTIONS:
Drug: Exendin-(9-39) — A physiological study to evaluate the role of GLP-1 signaling in glucose tolerance and insulin secretion
  Other Names: No other name for Exendin-(9-39)
  Arms: Exendin-(9-39)
Drug: Atropine — A physiological study to evaluate the effect of neural activation on insulin secretion and glucose metabolism
  Other Names: Atropine sulfate
  Arms: atropine
Drug: GLP-1 and GIP — A physiological study to evaluate the beta-cell sensitivity to different doses of exogenous gut hormones
  Other Names: No other names for GLP-1 and GIP.
  Arms: GLP-1 and GIP

SUMMARY:
RYGB (roux-en-y gastric bypass) has been reported to reverse type 2 diabetes (T2DM) immediately after surgery before any significant weight loss. In addition, a growing number of patients have been recognized with life-threatening hyperinsulinemic hypoglycemia several years following their surgery. While the mechanisms by which RYGB improves glucose metabolism or alters islet cell function in patients after RYGB are not understood, recent studies suggest that increased secretion of GI hormones, primarily glucagon-like peptide 1 (GLP-1), as well as alteration in neural activity may contribute to enhanced insulin secretion in general, and to a greater extent in patients with hypoglycemia. The proposed research is designed to address the role of RYGB on insulin secretion by evaluating the contribution of stimulatory factors (neural and GI hormone) on islet cell function and the islet cell responsiveness to the physiologic stimulatory factors, in RYGB patients with and without hypoglycemia and non-operated controls.

DETAILED DESCRIPTION:
RYGB (roux-en-y gastric bypass) has been reported to reverse type 2 diabetes (T2DM) immediately after surgery before any significant weight loss. In addition, a growing number of patients have been recognized with life-threatening hyperinsulinemic hypoglycemia several years following their surgery. While the mechanisms by which RYGB improves glucose metabolism or alters islet cell function in patients after RYGB are not understood, recent studies suggest that increased secretion of GI hormones, primarily glucagon-like peptide 1 (GLP-1), as well as alteration in neural activity may contribute to enhanced insulin secretion in general, and to a greater extent in patients with hypoglycemia. The proposed research is designed to address the role of RYGB on insulin secretion by evaluating the contribution of stimulatory factors (neural and GI hormone) on islet cell function and the islet cell responsiveness to the physiologic stimulatory factors, in RYGB patients with and without hypoglycemia and non-operated controls

ELIGIBILITY:
Inclusion Criteria:

* Hypoglycemic RYGB patients with documented blood glucose level <50 mg/dl
* Asymptomatic individuals with bariatric surgery
* Healthy non-surgical patients with no personal history of diabetes
* Subjects must physically be able to come to our clinical research center at Cedars-Sinai Medical Center

Exclusion Criteria:

* Active heart, lung, liver, gastrointestinal or kidney disease; unable to give informed consent; pregnancy; uncontrolled high blood pressure or high cholesterol; significant anemia (hemoglobin <11g/dL); prisoners or institutionalized individuals; type 2 diabetes melitis; development of any serious medical or psychiatric illness during recruitment or studies;
* RYGB patients will also be disqualified if they have gastric outlet obstruction or severe diarrhea
* Healthy non-surgical patients with personal history of diabetes

For administration of atropine, the following exclusions also apply:

* History of glaucoma
* Uncontrolled hypertension (any subjects with BP>140/90 and history of dyslipidemia
* Taking any medication that might interact with atropine and cannot be stopped will be excluded from the study)
* Myasthenia gravis
* Brain pathology
* Enlarged prostate in men

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-10; Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Gut hormones and neural signaling contribution to insulin secretion rate and glucose tolerance | Each study of the protocol is conducted up to seven hours with data collected at intervals specific to the individual study procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Marzieh Salehi, MD, MS, Principal Investigator — Marzieh Salehi
Locations (2):
- United States (2):
  - Texas Diabetes Institute - University Health System, San Antonio, Texas
  - South Texas Veterans Health Care System, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No